CLINICAL TRIAL: NCT04113200
Title: Gastric, Biochemical, Endocrine and Appetitive Responses to an Enterally Fed Alginate-containing Feed, Compared With an Alginate Free Feed
Brief Title: Comparison of an Alginate Containing Enteral Feed and an Alginate Free Enteral Feed.
Acronym: AlgiNG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Kaneka Corporation (Industry)
Responsible Party: Principal Investigator, Moira Taylor, Principal Investigator, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RGS129061
Record Dates: First submitted 2019-07-11; First posted 2019-10-02 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Enteral Nutrition

STUDY DESIGN:
Intervention Model Description: Participants will receive the control and intervention product according to randomised crossover design with a minimum washout period of 7 days.
Who Masked: Participant, Outcomes Assessor
Masking Description: On each study day, when the feed is administered, the Principle investigator (if present) and the research nurse administering the feed and obtaining blood samples are aware of which enteral feed will be given, but the MRI (magnetic resonance imaging) scanner, and researcher collecting outcome data will not be.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F+ALG (Experimental): An alginate containing feed: MerMed One (Kaneka Corporation). 300mls administered nasogastrically over one hour.
  Interventions: Dietary Supplement: MerMed One
- F-ALG (Other): A standard enteral feed commonly used in practice. Nutricomp Soy Fibre (B.Braun). 300mls administered nasogastrically over one hour.
  Interventions: Dietary Supplement: Nutricomp Soy Fibre

INTERVENTIONS:
Dietary Supplement: MerMed One — A 1 kcal per ml enteral feed containing an alginate.
  Arms: F+ALG
Dietary Supplement: Nutricomp Soy Fibre — A 1kcal per ml enteral feed not containing alginate.
  Arms: F-ALG

SUMMARY:
When patients cannot eat and drink enough a tube can be placed through their nostril, down the back of their throat into their stomach and used to give their nutrition as a liquid feed. One of the commonest problems when using this tube is regurgitation of feed up from the stomach (gastro- oesophageal reflux (GOR)), or liquid stools (diarrhoea). This can cause the patient discomfort, a higher risk of getting a skin or chest infection, and increase the risk that the feed is stopped.

The investigators intend to investigate, in twelve healthy young men, whether adding a form of dietary fibre (alginate) to the feed could reduce these symptoms (diarrhoea and GOR), hence ensuring patients are properly nourished and recover as quickly as possible from their illness, Each volunteer will come to the lab twice and will have a tube inserted into the stomach via the nose so that they can be given both feeds. Each time, the investigators will take repeated pictures of how the feed is passing through their gut using a non invasive technique called 'magnetic resonance imaging' (MRI), take blood samples to see how quickly the nutrition is absorbed into the blood, and measure how hungry they feel

DETAILED DESCRIPTION:
TRIAL / STUDY DESIGN Each participant will be required to attend a screening visit, a brief education visit re collecting dietary information, adhering to a standardised diet and faecal sample collection; two, approximately five hour, study visits with 7- 10 days between each visit; and a brief visit after each intervention day to return diet information and the faecal samples. Prior to the study visits they will be required to consume a standardised diet for four days, based on their usual intake with similar macronutrient composition to the feed. On each study visit they will be fed, via a nasogastric enteral tube, 300mls/ hour of one of two enteral feeds (total feed delivered 300mls). The gastric response will be measured using MRI scanning, the biochemical and endocrine response will be measured using arterialised venous blood samples, and the appetitive response will be measured using visual analogue scales, and direct measurement of food intake at an ad libitum test meal. Participants will continue to consume a standardised diet for 3 days after the delivery of the enteral feed. Faecal samples will be collected before and after the visit day, for pH measurement.

Ethical approval has been obtained from the Faculty of Medicine and Health Sciences Ethics Committee, University of Nottingham. All participants will provided informed, written consent.

ELIGIBILITY:
Inclusion Criteria:

* Non- smoking (non- vaping) males
* aged 18- 45 years
* body mass index (BMI) of 18.5-24.5kg/ m2 or a BMI of 24.5- 26kg/ m2
* a waist circumference of less than 94 cm.
* ability to give informed consent

Exclusion Criteria:

* A history of an acute illness, lasting more than a week, in the last six weeks;
* taking any medications for gastrointestinal disorders, including acid suppressants or anti-spasmodics,
* taking anti-depressants or symptoms of clinical depression (defined by a score >10 on the Beck Depression Inventory)
* taking medication for diabetes or having diabetes
* a history of substance abuse in the last six months;
* having any factors that preclude safe MRI;
* a history of gastrointestinal disorders, including Gastro Oesophgeal Reflux Disease, Irritable Bowel Syndrome, active peptic ulcer disease; having diabetes;
* previous surgery to the gastrointestinal or biliary systems;
* having characteristics of those with an eating disorders (defined by a score of more than 20 on the Eating Attitudes Test (EAT-26));
* having an allergy or intolerance to the ingredients in the enteral feeds, or the cheese and tomato pasta meal

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Small bowel water response to feeding | After four hours from baseline
  Area under the curve for small bowel water measured by MRI over four hours from baseline.

SECONDARY OUTCOMES:
Gastric volume relative to baseline | After four hours from baseline
  Area under the curve for gastric volume relative to baseline, measured by MRI for four hours from baseline.
Mean post feeding gastric emptying rate | Over four hours from baseline.
  Mean gastric emptying rate calculated from MRI images of gastric volume obtained over four hours from baseline.
Superior mesenteric blood flow | Over four hours from baseline.
  Mean superior mesenteric blood flow calculated from measurements over four hours from baseline.
Incremental area under the curve for arterialised whole blood glucose | Over four hours post baseline
  Incremental area under the curve for arterialised whole blood glucose will be calculated using samples collected at 10 minute intervals between baseline and four hours.
Incremental area under the curve for insulin | Over four hours from baseline
  Incremental area under the curve for insulin will be calculated using samples collected at 20 minute intervals between baseline and four hours.
Incremental area under the curve for PYY (Peptide YY) | Over four hours from baseline
  Incremental area under the curve for PYY will be calculated using samples collected at 20 minute intervals between baseline and four hours.
Incremental area under the curve for Gastric Inhibitory Polypeptide | Over four hours from baseline
  Incremental area under the curve for GIP will be calculated using samples collected at 20 minute intervals between baseline and four hours.
Incremental area under the curve for Glucagon-like peptide 1 (GLP- 1) | Over four hours from baseline
  Incremental area under the curve for GLP-1 will be calculated using samples collected at 20 minute intervals between baseline and four hours.
Incremental area under the curve for Ghrelin | Over four hours from baseline
  Incremental area under the curve for Ghrelin will be calculated using samples collected at 20 minute intervals between baseline and four hours.
Incremental area under the curve for composite satiety score | Over four hours from baseline
  Composite satiety score will be calculated using 100mm visual analogue score ratings of satiety, fullness, hunger and prospective food consumption collected every 30 minutes between baseline and four hours.
Weight of consumption of a pasta meal four hours and thirty minutes after baseline. | Four hours and thirty minutes post baseline.
  Weight of pasta consumed from a bowl refilled prior to being empty until participants feel comfortably full.
Change in Faecal pH from baseline | Comparison between sample obtained immediately before the enteral feeding day and samples obtained during the three days following the enteral feeding day.
  The difference between faecal pH pre feeding and post feeding will be compared.
Faecal consistency | Comparison between sample obtained immediately before the enteral feeding day and samples obtained during the three days following the enteral feeding day.
  Rating of consistency of faecal sample will be compared with rating of consistency post enteral feeding day.
Incremental area under the curve for gastric symptom scores rated using visual analogue scores. | Over four hours from baseline.
  Incremental area under the curve for gastric symptoms will be calculated using 100mm visual analogue score ratings obtained every half hour between baseline and four hours.

CONTACTS AND LOCATIONS:
Overall Officials: Moira Taylor, PhD, Principal Investigator — University of Nottingham
Locations (1):
- The University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised individual personal data will be shared, upon specific request from other researchers, for example, in order to undertake a meta analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When requested.
Access Criteria: On receipt of requests, data will be made accessible if agreed by both the University of Nottingham and Kaneka Corporation.